CLINICAL TRIAL: NCT06664411
Title: Polatuzumab Vedotin, Zanubrutinib, Rituximab, Lenalidomide and Prednisone in Previously Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Pola-ZR2P in Previously Untreated DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Associate Chief Physician, Associate Professor, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIME01
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; zanubrutinib; Rituximab; Lenalidomide; Prednisone; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pola-ZR2P (Experimental): Patients were treated by Pola-ZR2P as Induction Therapy
  Interventions: Drug: Polatuzumab Vedotin, Zanubrutinib, Rituximab, Lenalidomide and Prednisone as Induction Therapy

INTERVENTIONS:
Drug: Polatuzumab Vedotin, Zanubrutinib, Rituximab, Lenalidomide and Prednisone as Induction Therapy — Patients were treated by Polatuzumab Vedotin(1.8mg/kg iv qd d1), Zanubrutinib(160mg po bid d1-21), Rituximab(375mg/m2 iv qd d1), Lenalidomide(25mg po qd d1-14) and Prednisone(60mg/m2 po qd d1-5) as induction therapy
  Other Names: Pola-ZR2P

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of Pola-ZR2P as induction therapy in patients with DLBCL.

DETAILED DESCRIPTION:
The investigators will evaluate safety and efficacy of Pola-ZR2P as induction therapy in Previously Untreated Diffuse Large B-Cell Lymphoma. ORR(Overall response rate, progression-free survival (PFS), overall survival (OS), adverse events (AEs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Diffuse Large B Cell Lymphoma according World Health Organization (WHO) classification;
* Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted;
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements;
* Patient has not received chemotherapy previously.
* Anticipated life expectancy at least 3 months

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.
* Pregnant or lactating women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression was defined according to the Lugano Response Criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 years
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Overall Response Rate (ORR) | 1 year
  ORR was defined as the proportion of patients who achieved CR or PR

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, PhD, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China